CLINICAL TRIAL: NCT01039467
Title: Study of a Comparison of the Pacemaker Automatic Features in Reduction of Ventricular Pacing
Brief Title: A Comparison of the Pacemaker Automatic Features in Reduction of Ventricular Pacing
Acronym: COMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMPARE Study
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Bradycardia
Keywords: Managed Ventricular Pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Managed Ventricular Pacing (Active Comparator): Managed Ventricular Pacing group: programmed on
  Interventions: Device: Medtronic Adapta Dual Chamber Pacemaker
- Search AV+ (Active Comparator): Search AV+: programmed on
  Interventions: Device: Medtronic Adapta Dual Chamber Pacemaker

INTERVENTIONS:
Device: Medtronic Adapta Dual Chamber Pacemaker — Medtronic Adapta Dual Chamber Pacemaker

SUMMARY:
The COMPARE-Adapta study is a randomized, multi-center, prospective study conducted in China. The purpose of the study is to compare the ability of Search AV™+ and Managed Ventricular Pacing® (MVP®) to reduce ventricular pacing in dual chamber pacemaker-indicated patients. The COMPARE-Adapta study will also observe atrial fibrillation (AF) burden as demonstrated by Cardiac Compass® and the clinical profile Adapta® pacemaker patients.

DETAILED DESCRIPTION:
Recent studies suggest that chronic right ventricular pacing is associated with a variety of adverse effects in patients, particularly those with intact or intermittent atrioventricular (AV) conduction.

Medtronic Adapta® pacemakers include Managed Ventricular Pacing®, a pacing mode designed to promote intrinsic conduction, and also Search AV™+, a feature designed to reduce unnecessary ventricular pacing in patients with intact or intermittent AV conduction.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated study informed consent
* Class I or Class IIa pacemaker indication
* Geographically stable and available for follow-up at the center for the length of the study
* Age greater than 18
* To be implanted with Adapta dual chamber pacemaker

Exclusion Criteria:

* Unwillingness or inability to give written informed consent to participate in the Study
* Patient with a previously implanted pacemaker/Implantable Cardioverter-Defibrillator (ICD)/Cardiac Resynchronization Therapy (CRT) device
* Life expectancy of less than one year
* Patient has a mechanical tricuspid heart valve
* Medical conditions that preclude the testing requirement by the protocol or limit study participation
* Patient has persistent 3rd degree atrioventricular (AV) block
* Patient has persistent atrial fibrillation (AF)
* Patient has neurogenic syncope
* Patient has carotid sinus syndrome
* Patient has hypertrophic obstructive cardiomyopathy
* Inclusion in another clinical trial or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu Zhang, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (30):
- China (30):
  - 3rd Hospital of Beijing University, Beijing, Beijing Municipality
  - Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Fujian Province Hospital, Fuzhou, Fujian
  - 1st Hospital of Zhongshan Medical University, Guangzhou, Guangdong
  - 2nd Hospital of Zhongshan Medical University, Guangzhou, Guangdong
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - 1st Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Asian Heart Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Second Hospital, Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - 2nd Hospital of Jilin University, Changchun, Jilin
  - Liaoning Province People's Hospital, Shenyang, Liaoning
  - Affiliated Hospital of Qingdao Medical College, Qingdao, Shandong
  - Shanghai Huadong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Hospital, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xinjiang Automatic District Hospital, Ürümqi, Xinjiang
  - 1st Hospital of Kunming Medical College, Kunming, Yunnan
  - Yunnan Province 1st People's Hospital, Kunming, Yunnan
  - Yuxi People's Hospital, Yuxi, Yunnan
  - 1st Hospital of Medical College, Zhejiang University, Hangzhou, Zhejiang
  - 2nd Hospital of Medical College, Zhejiang University, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Shanghai First People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: 18 JUN 2009 to 15 MAR 2010.
Pre-assignment Details: 6 patients withdrawn from study pre-randomization for not meeting inclusion/exclusion criteria.
Groups:
- Managed Ventricular Pacing (MVP): Managed Ventricular Pacing (MVP) used in dual chamber pacemaker
- Search AV+: Search AV+ used in dual chamber pacemaker
Period: Overall Study
Arm/Group | Managed Ventricular Pacing (MVP) | Search AV+
Started | 196 | 189
Completed | 156 | 140
Not Completed | 40 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Managed Ventricular Pacing (MVP) | Search AV+ | Total
Number analyzed (Participants) | 196 | 189 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.87 (10.35) | 70.71 (9.89) | 70.28 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 81 | 174
  Male | 103 | 108 | 211
Region of Enrollment [Number; unit: participants]
  China | 196 | 189 | 385

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decreased Percent of Ventricular Pacing Compared to MVP Using Search AV+
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with %VP data available.
Measure: Count of Participants; unit: Participants
Groups:
- Managed Ventricular Pacing: Managed Ventricular Pacing (MVP)
- Search AV+: Search AV+ (SAV+)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 167 | 163
Participants | 1 | 4
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent of Ventricular Pacing
Time Frame: 12 months post-implantation
Population: all participants who completed the 12 months visit with %VP data available.
Measure: Median (Standard Deviation); unit: percent of ventricular pacing (%VP)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 156 | 140
percent of ventricular pacing (%VP) | 0.40 (31.46) | 2.95 (40.05)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Reduced Percent of Atrial Fibrillation (AF) Burden 1-month Post-Implant
Description: To compare the ability of Search AV™+ and Managed Ventricular Pacing® (MVP®) to reduce ventricular pacing in dual chamber pacemaker-indicated patients by measuring the percent burden of atrial fibrillation (AF) burden as demonstrated by Cardiac Compass® and the clinical profile Adapta® pacemaker patients.
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with
  %AT/AF burden data available.
Measure: Median (Standard Deviation); unit: Percentage of decreasedAT/AF burden
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 37 | 35
Percentage of decreasedAT/AF burden | 1.40 (20.27) | 0.50 (25.43)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p = 0.833, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Percent of Ventricular Pacing
Time Frame: from 1 month to 12 months post-implantation
Population: all participants who completed the 12 months visit with %VP data available.
Measure: Median (Standard Deviation); unit: percent of ventricular pacing (%VP)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 141 | 129
percent of ventricular pacing (%VP) | -0.10 (20.20) | 0.00 (20.18)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p = 0.265, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Percent Ventricular Pacing Reduced to Lower Levels (<10%VP)
Time Frame: 1 month post-implantation
Population: all participants who completed the 12 months visit with %VP data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 167 | 163
Participants | 132 | 91
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p < 0.0001, Chi-squared

6. Secondary Outcome: Number of Participants With Decreased Percent Ventricular Pacing Stratified by Baseline Atrioventricular Block Status (No AVB - nAVB)
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with %VP data available.
Measure: Count of Participants; unit: Participants
Groups:
- No AV Block: Patients with no atrioventricular block
- nAVB: Patients with atrioventricular block
Arm/Group | No AV Block | nAVB
Number analyzed (Participants) | 105 | 110
Participants | 1 | 1
Statistical Analysis 1: Comparison: No AV Block vs nAVB; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent of Ventricular Pacing Stratified by Baseline AV Block Status (1st Degree - 1AVB)
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with %VP data available.
Measure: Median (Standard Deviation); unit: percent of ventricular pacing (%VP)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 18 | 10
percent of ventricular pacing (%VP) | 1.50 (23.65) | 21.80 (41.00)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p = 0.0008, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percent of Ventricular Pacing Stratified by Baseline AV Block Status (2nd Degree Type I & II - 2AVB)
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with %VP data available.
Measure: Median (Standard Deviation); unit: percent of ventricular pacing (%VP)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 31 | 33
percent of ventricular pacing (%VP) | 21.40 (39.16) | 80.60 (44.03)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing vs Search AV+; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Percent of Ventricular Pacing Stratified by Baseline AV Block Status (3rd Degree Episodic - e3AVB)
Time Frame: 1 month post-implantation
Population: all participants who completed the 1 month visit with %VP data available.
Measure: Median (Standard Deviation); unit: percent of ventricular pacing (%VP)
Arm/Group | Managed Ventricular Pacing | Search AV+
Number analyzed (Participants) | 13 | 10
percent of ventricular pacing (%VP) | 79.20 (44.68) | 22.45 (47.13)
Statistical Analysis 1: Comparison: Managed Ventricular Pacing; Test type: Superiority or Other; p = 0.493, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Managed Ventricular Pacing | Search AV+
Serious Adverse Events (participants affected / at risk) | 2/196 | 7/189
Other Adverse Events (participants affected / at risk) | 2/196 | 3/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Managed Ventricular Pacing (N=196) | Search AV+ (N=189)
Death (unknown reason) (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (CHD) (General disorders) | 0 (0) | 2 (2)
Non-cardiac death (cancer) (General disorders) | 0 (0) | 2 (2)
Non-cardiac death (cerebrovascular accident） (General disorders) | 0 (0) | 1 (1)
Pocket infection (Infections and infestations) | 1 (1) | 0 (0)
Dislodgement of RV lead and reposition of the lead (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Managed Ventricular Pacing (N=196) | Search AV+ (N=189)
dizziness (Nervous system disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No